CLINICAL TRIAL: NCT04786041
Title: Lockdown With a Price- the Impact of COVID-19 Pandemic on the Incidence and Outcome of Complicated Appendicitis
Brief Title: the Impact of COVID-19 Pandemic on the Incidence and Outcome of Complicated Appendicitis
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yaron rudnicki, attending surgeon - surgical ward B, Meir medical center, Meir Medical Center
Other Study IDs: MMC-0223-20
Record Dates: First submitted 2021-03-05; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Appendicitis
Keywords: COVID19; appendicitis; laparoscopy
MeSH Terms: conditions — COVID-19; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- underwent Appendectomy during march-april of 2019: all patients who underwent Appendectomy during the period of march-april of 2019
  Interventions: Procedure: laparoscopic appendectomy
- underwent Appendectomy during march-april of 2020 (during covid pandemic): all patients who underwent Appendectomy during the period of march-april of 2020 (during the COVID19 pandemic lockdown)
  Interventions: Procedure: laparoscopic appendectomy

INTERVENTIONS:
Procedure: laparoscopic appendectomy — laparoscopic appendectomy
  Other Names: abscess drainage; consevative treatment

SUMMARY:
During the COVID-19 pandemic, we noticed a rise in complicated appendicitis cases presenting to our medical center. We collected objective data on all patients admitted to the surgical department with appendicitis during February 2020 - March 2020 compared to the same 2 month period in 2019, to understand the pandemic's affect on the rate of complications of acute appendicitis.

DETAILED DESCRIPTION:
Coronavirus pandemic (COVID-19) first broke out in Wuhan and Hubei China during december 2019. On 30 January, WHO declared it a Public Health Emergency of International Concern (PHEIC) .

Currently, the number of cases worldwide stands stands at more than 76 million confirmed cases according to the World Health Organization (WHO) records. First documented case in Israel was reported on 21st of february 2020.

During the months of February and April, due to continued rise in confirmed cases, rigid "stay at home" restrictions were issued. These restrictions have had a significant effect on daily life. Under these new "stay at home" policies, many aspects of everyday life were greatly diminished and restricted under threat of heavy fines. This effect also extends to reduction in healthcare seeking. decline in emergency department (ED) visits was reported. A drop in routine cancer screening appointments was reported.

Delayed healthcare seeking also had an affect on the severity of various medical conditions on presentation. fear of the COVID-19 pandemic may have resulted in delayed diagnosis, and therefore higher complication rates in common medical conditions.

acute appendicitis (AA) is among the most common causes of lower abdominal pain leading patients to attend the emergency department. As such, AA could serve as a good indicator for the possible effect that the fear of the COVID-19 pandemic had on patients tendency for late diagnosis and complication rate.

Gomes Laparoscopic Grading System of AA, classifies appendicitis into five laparoscopic grades according to gross morphologic findings during surgical laparoscopy. grades 1 and 2 regarded as non-complicated appendicitis, while grades 3, 4 and 5 regarded as complicated appendicitis.

Following the restrictions imposed during the COVID-19 pandemic, we noticed a rise in complicated appendicitis cases presenting to our medical center. We collected objective data on all patients admitted to the surgical department with appendicitis during February 2020 - March 2020 compared to the same 2 month period in 2019. Data such as the time period from onset of symptoms to presenting to the ED, inflammatory markers, complicated appendicitis (if any), type of complication, post operative complications. We aim to assess whether the "stay at home" restrictions had any adverse effects on severity or outcomes of AA.

ELIGIBILITY:
Inclusion Criteria:

* appendicitis

Exclusion Criteria:

* any other diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients who underwent appendectomy in meir medical center, during the study period
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
complicated appendicitis | 30 days
  any complication during surgery or post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rudnicki, MD, Study Director — Meir medical center, surgical ward B.; Yaron Rudnicki, MD, Principal Investigator — Meir medical center, surgical ward B.
Locations (1):
- Meir medical center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rudnicki Y, Soback H, Mekiten O, Lifshiz G, Avital S. The impact of COVID-19 pandemic lockdown on the incidence and outcome of complicated appendicitis. Surg Endosc. 2022 May;36(5):3460-3466. doi: 10.1007/s00464-021-08667-9. Epub 2021 Jul 26. PMID 34312724